CLINICAL TRIAL: NCT05302154
Title: Virtual Reality as a Distraction Technique in Paediatric Dental Care, Assessment of Resulting Effects on Patient Anxiety, Pain and Behaviour
Brief Title: Effect of Virtual Reality on Dental Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Collaborators: Istanbul Technical University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 119S618
Record Dates: First submitted 2022-01-04; First posted 2022-03-31 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Behavior, Child
Keywords: behaviour management techniques; children; distraction; virtual reality
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Behavioral: Behavioral guidance Other: Pain assessment Other: Dental anxiety assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard treatment group (Active Comparator): Dental treatment is carried out with tell-show-do technique as a behavioural guidance technique.
  Interventions: Behavioral: Distraction by dentist
- Cartoon movie- passive distraction group (Experimental): Dental treatment is carried out with showing cartoon movie as a passive distraction during the treatment.
  Interventions: Behavioral: Distraction by cartoon movie
- VR-active distraction group (Experimental): The active distraction group is treated while wearing the VR headset and interacting with the designed application.
  Interventions: Behavioral: Distraction by virtual reality glasses

INTERVENTIONS:
Behavioral: Distraction by dentist — Basic behavior orientation techniques (tell-show-do) is applied by the dentist during the treatment.
  Arms: Standard treatment group
Behavioral: Distraction by cartoon movie — Children watch cartoons on a screen mounted dental unit during the treatment.
  Arms: Cartoon movie- passive distraction group
Behavioral: Distraction by virtual reality glasses — During the treatment visual and auditory stimuli provide information about treatment to the patient with the help of avatars (characters) and environmental elements placed within the VRG application. In a vivid dentist room, the explanatory introduction part takes place while the movies are watched in a fairy world or a futuristic world to separate the user from the actual location and context. The application was designed to function in such a way as not to require outside intervention. From start to finish, the application interacts with the user through gaze selection and head tracking mechanisms. The avatar characters provide information related to the dental treatment in a joyful manner. Gamification elements such as gaining stars and collecting rewards have been used to keep the patient engaged. Motion blur feature ensures the patient to keep head still as sudden movements are dangerous and undesired by the dentist during the treatment.
  Arms: VR-active distraction group

SUMMARY:
The aim of this study is to reduce dental anxiety in children by using virtual reality glasses (VRG) with a special content and innovative interactive methods, to determine the level of stress experienced by patients during dental treatment and to ease the workload of dentists.

Within the scope of the study, the participants being examined are in a controlled manner from the practice environment. They are attached a VRG and headphones throughout the treatment. With the help of VRG, it is ensured that participants are ready for the treatment. During the treatment, the participant's focus is on various contents in terms of spectacles. Contents include visual (video surveillance) and auditory stimuli (listening to music). They also provide information about treatment to the patient with the help of avatars (characters) and environmental elements that are placed into the VRG application. In addition, dental anxiety is reduced by the fun contents. The goal is to increase the rate of dental treatment success in child patients.

The effectiveness of virtual reality system is tested by comparing evaluation metrics of three groups of children. In the first group, the dentist carries out the treatment alone. In the second group participants watch cartoons on a screen mounted dental unit during the treatment. In the third group, dental treatment is carried out with VRG. In the course of these experiments, the effects of VRG on dental treatment (vital pulpotomy and dental filling) that require local anesthesia is examined in order to measure the effects of VRG on the level of stress on dental treatment.

Corresponding measures are; (1) the child's anxiety; (2) the child's pain perception during local anaesthesia and treatment; (3) the child's cooperation and general behaviour. The outcomes of the child's anxiety, pain perception, cooperation and general behaviour for three groups were evaluated by statistical analysis.

DETAILED DESCRIPTION:
The study is being carried out in Istanbul University Department of Pedodontics, period between March 2021 - December 2021 following the ethics committee approval 2018/5. Patient parents are informed about the study following the initial dental examination of the patient and the written informed consents are obtained from parents of all participants included in the study.

In this randomised parallel clinical study, the sample consisted of 90 children aged between 6-10 years old who applied for routine dental care in paediatric clinic.

Randomization Children are evaluated by the same dentist during the first examination with Frankl Behavior Rating Scale (FBRS) according to their behavioral attitudes and listed by numbers according to the order of application. Participants who do not come to the treatment appointment are recruited again. The volunteers in the top 30 on the list were recruited to Group I (GI), the next 30 volunteers to Group II (GII), and the last group of 30 volunteers to Group III (GIII).

Group I. Dental treatment is carried out using tell-show-do. Group II. Dental treatment is carried out with showing cartoon movie as a passive distraction.

Group III. The active distraction group is treated while wearing the VR headset and interacting with the designed application.

Study Procedure:

The success of the proposed approach is analyzed by the researcher observing the treatment session child's behaviours and physiological data. Pre-operative pulse rate is got from a pulse oximeter to evaluate the child's anxiety objectively. Children's Fear Survey Schedule-Dental Subscale is applied before the beginning of each visit to evaluate the child's subjective anxiety. In addition, FBRS is applied by the dentist. Video recordings are used to measure behavioral responses of the child before the treatment. Facial Image Scale is applied to children before the treatment to measure the pain perception of the children.

During the treatment, pulse rate is got from a pulse oximeter starting from the local anaesthesia application just before, during and after the treatment of local anesthesia.

The details of the treatment to be applied is as follows: Local anaesthesia application, the intraoral procedure with a high-speed rotary instrument, matrix application, restorative treatment (etch/adhesive application/polymerase/composite application with light-curing), finishing.

As soon as the treatment is completed, post-operative pulse rate, Facial Image Scale, Children's Fear Survey Schedule, FBRS are repeated. Moreover at the end of the dental treatment, children are asked whether they are willing to use VR in their next appointment. The answers given to this question are evaluated in 5 stages between "I would never want to" and "I would like it very much". Also dental chair sitting time of the participant during the procedure is recorded in the experimental and control groups.

The anticipated treatment time is determined as 30 minutes. The treatments are planned to be completed in a single session under local anesthesia. Parents are not allowed be with their children during the treatment according to the routine clinical procedure. A fixed camera which is placed in front of the child is used to record the sessions. Facial and body expressions records are evaluated with FBRS.

Basic behavior orientation techniques (tell-show-do, positive encouragement) is applied by the dentist during the treatment of the first group. According to a study in Turkey published in 2019, the most preferred movies were "Super Wings" for boys and "Frozen" for girls. Therefore, these movies are used in group II and group III. VR headset are used during the treatment of the third group. In a vivid dentist room, the explanatory introduction part takes place while the movies are watched in a fairy world or a futuristic world to take the user away from the real world. Specially created animations have enhanced the virtual environment. The application is designed to function in a way not requiring any intervention. From start to the end, the application interacts with the patient using gaze selection and head tracking mechanisms. The avatar characters provide information related to the dental treatment in a joyful manner. Gamification elements such as gaining stars and collecting rewards have been used to keep the patient engaged. Motion blur feature ensures the patient to keep his head still as sudden movements are supposed to be dangerous and undesired by the dentist during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Systemically and mentally healthy patients without any previous dental treatment experience,
* Children who required pulpotomy in lower primary molars under local anaesthesia.

Exclusion Criteria:

* Systemic disease,
* Mental and cognitive disorders, visual and auditory disabilities.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Child's behaviour assessment (subjective) Child's pain assessment (subjective) | 1 year
  According to the The Frankl Behavior Rating Scale, the child's attitude towards treatment is divided into 4 groups and scored between 1-4 meaning: 1 point absolutely negative (child refuses treatment, strong fear and crying), 2 points negative (reluctant to accept treatment), 3 points positive (child accepts treatment, but is cowardly and timid) 4 points absolutely positive (compatible with pediatric dentist).

SECONDARY OUTCOMES:
Child's anxiety assessment (objective) | 1 year
  Heart rate is used to determine the anxiety levels of all treated children at certain critical moments of the treatment being. Significant differences in heart rate is compared between groups.
Child's anxiety assessment (subjective) | 1 year
  Children's Fear Survey Schedule-Dental Subscale consists of 15 questions covering different aspects of dental treatment. It was done by asking children to score from 1 (not at all) to 5 (extremely scared) for each question (1 = Not scared at all, 2 = Slightly scared, 3 = A little scared, 4 = Very scared, 5 = Extremely scared). All scores are added together and the total score is obtained between 15 and 75. 15-31 points indicate low level, 32-38 points to moderate, and 39 and above to indicate high level of anxiety. 5 minutes after the end of the dental treatment, children are asked whether they are willing to use VR in their next appointment. The answers given to this question are evaluated in 5 stages between "I would never want to" and "I would like it very much".
Child's pain assessment (subjective) | 1 year
  Facial Image Scale is aimed to measure the pain perception of the child during dental treatment. Subjective responses from children before and after dental treatment is evaluated with five different facial expressions ranging from "very happy" (1) to "very unhappy" (5). With this questionnaire, it is planned to measure the pain perception of the children and make a comparison between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Elif B Tuna Ince, Prof., Study Director — Department of Pedodontics, Faculty of Dentistry, Istanbul University
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No